CLINICAL TRIAL: NCT02089984
Title: Web Based Therapist Training on Cognitive Behavior Therapy for Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Psychological Consultation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth A. Kobak, Ph.D., Owner, Center for Psychological Consultation
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R44MH086951 (NIH); R44MH086951 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Anxiety Disorders; Obsessive Compulsive Disorder; PTSD
Keywords: Cognitive Behavior Therapy; On-line training
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-Based Training (Experimental): On-line tutorial followed by live remote training via videoconferencing
  Interventions: Behavioral: Internet Based CBT Training

INTERVENTIONS:
Behavioral: Internet Based CBT Training

SUMMARY:
Anxiety disorders are a major public health concern, having a profound impact on functioning, causing significant disability, loss of productivity and suffering. Effective treatments exist for these disorders, but few clinicians are trained in these methods. This project attempts to remedy this shortcoming by using web-based tools to facilitate access to this training, thus increasing the number of available therapists in order to help meet this unmet need.

DETAILED DESCRIPTION:
The need for evidence-based mental health treatments i.e., 'treatment based on the best available science or research evidence', has been stressed from scientific, ethical, and economic perspectives. While empirical evidence supports both the efficacy and effectiveness of cognitive behavior therapy (CBT) for anxiety disorders, the demand for clinicians trained in these approaches far exceeds the supply. A major reason for this is the lack of trained cognitive behavior therapists. New technologies provide the opportunity to both facilitate accessibility to this specialized training by mental health professionals and to improve the quality of this training. Recent research has found that training clinicians using these new web-based technologies is highly effective, can significantly improve skills, and has significant advantages over traditional training programs. The long term goal of this project is to increase the number of available mental health professionals trained in cognitive behavior therapy for anxiety disorders by developing a set of web-based training tools enabling the widespread dissemination of this training. In Phase I the investigators developed a prototype online tutorial covering some core CBT principles and a Social Anxiety Disorder module. The investigators also tested the feasibility of live remote training through videoconferencing. In phase II investigators will expand the tutorial to include a comprehensive review of CBT principles and techniques and expand modules to include the full spectrum of anxiety and anxiety-related disorders (i.e., Obsessive Compulsive Disorder, Panic Disorder, Generalized Anxiety Disorder, Posttraumatic Stress Disorder and Social Anxiety Disorder). Investigators will also evaluate the efficacy of live remote training in improving clinical skills. A cohort of 50 clinicians from diverse educational and professional backgrounds will be recruited. Improvement in trainees' conceptual knowledge will be evaluated pre and post tutorial, and improvement in trainees' clinical skills in applying the CBT concepts will be evaluated by blind ratings of clinical adherence and competence at three time points: before on-line training, and before and after videoconference training. User satisfaction with both the on-line tutorial and the videoconference training will also be evaluated. Impact of training on post-training patient outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians are eligible for this therapist training study if they are a licensed health care professional or are currently in a counseling related graduate training program

Exclusion Criteria:

* None, except for above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | after completion of tutorial, an expected average of 2 weeks
  User satisfaction with the technical aspects of the tutorial was assessed using the ratings on the System Usability Scale (SUS), a reliable, well-validated 10-item scale designed to evaluate the usability and user satisfaction with web-based applications and other technologies.
CBT Concepts | After completing the on line tutorial, an expected average of two weeks
  Improvement in trainees' knowledge of CBT concepts will be evaluated using a 38-item pre and post test of the items covering the tutorial content.

SECONDARY OUTCOMES:
Yale Adherence and Competence Scale (YACS) | At day 0 (baseline) (i.e., priot to any training), and after completing the on line tutorial (an expected average of two weeks), and after completing the appled training (an exected average of 8 weeks).
  The Yale Adherence and Competence Scale (YACS) is a well-validated, scale for rating therapist adherence and competence in delivering cognitive behavioral treatments. It has been used as an outcome measure in several studies evaluating the effectiveness of different CBT rater training approaches . Therapist competence in administering specific CBT techniques is evaluated on a scale ranging from 1 (very poor) to 7 (excellent).
User Satisfaction Questionnaire | After completing the on line tutorial (an expected average of 2 weeks)
  This scale evaluates how well subjects liked the clinical content of the on-line tutorial. It contains 14 statements, each of which are rated on a 4-point scale (strongly agree, agree, disagree, strongly disagree), and covers several dimensions of the user experience . The scale ranges from 15 to 60, and has good internal consistency reliability (Cronbach's Alpha =.90, Phase I study results). An overall mean score of 45 (i.e., an average score of 3 ("agree" on all items)) is considered adequate to demonstrate acceptable user satisfaction with the clinical content.

OTHER OUTCOMES:
GAD-7 | Weekly for 8 weeks of patient treatment, post training
  The GAD-7 is a well-validated self-report scale originally developed as a brief measure of GAD. It has since been validated as measure of anxiety across the domain of anxiety disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Telepsychology, Madison, Wisconsin, United States

REFERENCES:
- [Background] Kobak KA, Craske MG, Rose RD, Wolitsky-Taylor K. Web-based therapist training on cognitive behavior therapy for anxiety disorders: a pilot study. Psychotherapy (Chic). 2013 Jun;50(2):235-47. doi: 10.1037/a0030568. Epub 2013 Feb 11. PMID 23398031